CLINICAL TRIAL: NCT00001464
Title: Effect of Hypoxia and Smoking on Oxidation of Proteins and Nucleic Acids in Human Volunteers
Brief Title: Effect of High Levels of Oxygen and Smoking on the Lungs in Human Volunteers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950167; 95-H-0167
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
Keywords: Oxygen; Bronchoalveolar Lavage; DNA Repair; Carbonyl Groups; Serum; Human Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group 1: Smokers exposed to oxygen

SUMMARY:
Patients with lung disease experiencing difficulty breathing can be treated with oxygen therapy. This involves the delivery of "extra" oxygen by a face-mask or through small tubes placed in the nose called nasal prongs. This extra oxygen can have concentrations as high as 100% pure oxygen. The concentration of oxygen in normal air is only 21%. The high concentration of oxygen can help to provide enough oxygen for all of the organs in the body. Unfortunately, breathing 100% oxygen for long periods of time can cause changes in the lungs, which are potentially harmful. Researchers believe that by lowering the concentration of oxygen therapy to 40% patients can receive it for longer periods of time without the risk of side effects.

This study is designed to evaluate the effects of oxygen therapy at 100% and 40% for 12 18 hours on the lungs of normal volunteers. Results of this study will help to determine if levels of oxygen therapy currently accepted as being "safe" may actually be damaging to the lungs.

DETAILED DESCRIPTION:
Stress such as high oxygen or inflammation can result in damage to proteins by processes such as oxidation or alternative regulation of signaling pathways by post-translational modification of proteins (e.g., phosphorylation). Delivery of oxygen in high concentrations to the lungs can result in damage, which is mediated in large part by reactive oxygen species. Inflammation can result in activation of intracellular signaling pathways. This study will evaluate modification of proteins and nucleic acids in bronchoalveolar lavage fluid, bronchial epithelial cells, and peripheral blood of individuals exposed to oxygen or who are smokers. In doing so, it will determine the effects of hyperoxia or inflammation on the lung.

ELIGIBILITY:
* INCLUSION CRITERIA:

History - good overall health without history of recent (within 3 months) acute disease;

Physical examination within normal limits;

Laboratory evaluation; including complete blood count (CBC), serum electrolyte determinations, clotting times, chest x-ray, pulmonary function testing, and an electrocardiogram (EKG) - within normal limits;

Non-smokers defined as having never smoked or not smoked in the past 2 years;

Smokers defined as moderate (1 pack per day for 3+ years) or heavy (1-2 packs for 10+ years);

Subjects must be willing to make the time commitment necessary for the study.

EXCLUSION CRITERIA:

Any study subject who does not fulfill the criteria for eligibility.

Individuals with a history of allergy or adverse reactions to atropine or any local anesthetic;

Individuals testing positive for the human immunodeficiency virus or hepatitis virus;

Individuals on chronic medications or currently receiving medications;

Pregnant or lactating individuals, since the effects of hyperoxia on the fetus are unclear.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals exposed to oxygen or who are smokers.@@@
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 1995-08-22 (Actual); Primary Completion 2007-07-10 (Actual); Study Completion 2007-07-10 (Actual)

PRIMARY OUTCOMES:
To determine whether hyperoxia of relatively limited duration (up to l8 hrs) is associated with oxidation of proteins and nucleic acids in lung cells. | 1 week
  To determine whether hyperoxia of relatively limited duration (up to l8 hrs) is associated with oxidation of proteins and nucleic acids in lung cells.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Deneke SM, Fanburg BL. Normobaric oxygen toxicity of the lung. N Engl J Med. 1980 Jul 10;303(2):76-86. doi: 10.1056/NEJM198007103030204. No abstract available. PMID 6247652
- [Background] Erzurum SC, Danel C, Gillissen A, Chu CS, Trapnell BC, Crystal RG. In vivo antioxidant gene expression in human airway epithelium of normal individuals exposed to 100% O2. J Appl Physiol (1985). 1993 Sep;75(3):1256-62. doi: 10.1152/jappl.1993.75.3.1256. PMID 8226538
- [Background] Davis WB, Rennard SI, Bitterman PB, Crystal RG. Pulmonary oxygen toxicity. Early reversible changes in human alveolar structures induced by hyperoxia. N Engl J Med. 1983 Oct 13;309(15):878-83. doi: 10.1056/NEJM198310133091502. PMID 6888481
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1995-H-0167.html